CLINICAL TRIAL: NCT00793273
Title: Evaluation of Glycaemic Control After Initiation of Levemir® in Patients With Type 2 Diabetes Mellitus and Time Period Between Diagnosis of Type 2 Diabetes Mellitus and Insulin Initiation.
Brief Title: Observational Study to Observe the Efficacy of Levemir® (Insulin Detemir) in Patients With Type 2 Diabetes.
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3694
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Effectiveness and safety data collection in connection with the use of the drug Levemir® in daily clinical practice
  Other Names: Levemir®; NN304

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to observe the efficacy of Levemir® treatment in patients with type 2 diabetes in everyday clinical practice in Switzerland. Furthermore the time period between diagnosis of type 2 diabetes and insulin initiation is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus
* Insulin-naive or currently treated with another basal insulin
* Inclusion of patients at the discretion of the treating physician after the decision to prescribe Levemir®

Exclusion Criteria:

* Type 1 diabetes mellitus
* Patients treated with short acting or with premix insulin
* Women who are pregnant, breast feeding or have the intention to become pregnant
* Known or suspected allergy to the study product or related product
* Any exclusion criteria according to the Swiss Levemir® SPC (Summary of Product Characteristics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from general practice setting who have been deemed appropriate to receive Levemir® as part of routine out-patient care by the prescribing physician.
Sampling Method: Probability Sample
Enrollment: 1074 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c of treatment | after 12 to 16 weeks
Change in FPG (fasting plasma glucose) of treatment | after 12 to 16 weeks

SECONDARY OUTCOMES:
Occurrence of adverse events | after 12 to 16 weeks
Insulin dose and concomitant oral antidiabetic medication time period between diagnosis of type 2 diabetes and insulin initiation | after 12 to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Zurich, Oerlikon, Switzerland

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com